CLINICAL TRIAL: NCT04742439
Title: Testing the Effects of Individualized and 4mA tDCS
Brief Title: Individualizing tDCS Dose
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We currently do not have the time to pursue this research given other ongoing projects. If we restart this project, we will submit a new ClinicalTrials record for the protocol. Thank you.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kevin Caulfield, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 00104712; P2CHD086844 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: tDCS; Motor Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham transcranial direct current stimulation
- Individualized stimulation (Experimental)
  Interventions: Device: Individualized transcranial direct current stimulation
- 2mA stimulation (Experimental)
  Interventions: Device: 2mA transcranial direct current stimulation
- 4mA stimulation (Experimental)
  Interventions: Device: 4mA transcranial direct current stimulation

INTERVENTIONS:
Device: Sham transcranial direct current stimulation — Participants will receive 30 seconds of ramp up and down stimulation at the start and end of the 20 minute stimulation period.
  Arms: Sham stimulation
Device: Individualized transcranial direct current stimulation — Participants will receive 20 minutes of transcranial direct current stimulation (tDCS) at the individualized dose (maximum of 4mA).
  Arms: Individualized stimulation
Device: 2mA transcranial direct current stimulation — Participants will receive 20 minutes of transcranial direct current stimulation (tDCS) at a 2mA dose.
  Arms: 2mA stimulation
Device: 4mA transcranial direct current stimulation — Participants will receive 20 minutes of transcranial direct current stimulation (tDCS) at a 4mA dose.
  Arms: 4mA stimulation

SUMMARY:
Transcranial direct current stimulation (tDCS) is a noninvasive method of modulating brain activity and has therapeutic potential in many neurological and psychiatric conditions. However, unlike every current FDA-approved form of brain stimulation, there is no method of individualizing stimulation dose. In this study, a method of individualizing tDCS dose on behavioral outcomes and whether this could help to improve the consistency and magnitude of the stimulation effects will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers or chronic stroke participants (at least 6 months prior to the study)
* No history of epilepsy
* No metal in the body
* No contraindications for TMS or MRI scanning
* Right handed
* Ability to find motor hotspot and acquire motor evoked potentials

Exclusion Criteria:

* Metal in the body
* History of epilepsy or claustrophobia
* Alcohol or substance abuse or dependence
* Current treatment for any psychiatric conditions (pharmacological or otherwise)
* Pregnant or actively breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Motor Evoked Potential Variance | Baseline and post-stimulation (20 minutes apart)
  MEP variance is measured by single pulses of transcranial magnetic stimulation and contralateral hand electrodes.
Difference in Motor Evoked Potential Amplitudes from 4mA and 2mA Stimulation | Baseline and post-stimulation (20 minutes apart)
  MEP amplitude is measured by single pulses of transcranial magnetic stimulation and contralateral hand electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04742439/ICF_000.pdf